CLINICAL TRIAL: NCT03646552
Title: Feasibility Study - Whether the Administration of the Dronabinol and PEA May Act as a Therapy for Obstructive Sleep Apnea
Brief Title: A Study to Examine the Efficacy of a Therapeutic THX-110 for Obstructive Sleep Apnea
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Neurothera Labs Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0079-17-ASMC
Record Dates: First submitted 2018-08-05; First posted 2018-08-24 (Actual); Last update posted 2018-08-24 (Actual); Status verified 2018-08

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- THX-110 (Experimental): All participants will be titrated up on THX-110 (Dronabinol) dose during the first week of the trial (2.5mg Dronabinol for 3 days, 5mg Dronabinol for 3 days to 7.5mg Dronabinol for 3 days and finally increasing to 10mg for the remainder of the trial). Dronabinol will only be increased if the subject is tolerating the previous dose of Dronabinol and the Dronabinol may be reduced based on patient side-effects. Participants will be receiving 800mg PEA concomitantly.
  Interventions: Drug: THX-110

INTERVENTIONS:
Drug: THX-110 — Participants will receive THX-110 in the following regimen:
  Dronabinol will be slowly titrated in the first 10 days of the study and PEA will be given in a constant dose of 800mg per day for the entire duration of the study.
  Patients will be followed for a total of 30 days.

SUMMARY:
This is a sponsored proof of concept study with the purpose to examine the safety, tolerability and feasibility of THX-110 (Dronabinol (synthetic Δ9-THC) and PEA) for the treatment of adults with Obstructive Sleep Apnea.

DETAILED DESCRIPTION:
This is a 30-day sponsor-initiated, open-label trial of the therapeutic treatment THX-110 (a combination of Dronabinol and PEA) in 30 adults with Obstructive Sleep Apnea (OSA). Participants will receive THX-110 for the duration of the trial. The goal for this pilot study is to provide initial safety, feasibility and tolerability data on THX-110 in an OSA population.

ELIGIBILITY:
Inclusion Criteria:

* OSA diagnosis; OSA severity AHI: 15-30
* Population aged 20-65
* Gender: Males and Females
* BMI < 30
* OSA patients that cannot tolerate CPAP
* OSA patients who use CPAP will not use the device during the entire duration of the study

Exclusion Criteria:

* Minors
* Severity of OSA outside the determined boundaries
* Pregnancy
* BMI > 30
* Medical history of narcotic dependency

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-06-04 (Actual); Primary Completion 2019-04 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
A Significant Change in AHI Index | 30 days
  A significant change in AHI index, which assesses the quality of sleep before and after the treatment.
  The AHI is the number of apneas or hypopneas recorded during the study per hour of sleep. It is generally expressed as the number of events per hour. Based on the AHI, the severity of OSA is classified as follows:
  None/Minimal: AHI < 5 per hour Mild: AHI ≥ 5, but < 15 per hour Moderate: AHI ≥ 15, but < 30 per hour Severe: AHI ≥ 30 per hour

SECONDARY OUTCOMES:
A Change in Oxygen Desaturation Index (ODI) | 30 days
  A change in oxygen desaturation index (ODI) before and after the treatment
  ODI is the hourly average number of desaturation episodes, which are defined as at least 4% decrease in saturation from the average saturation in the preceding 120 seconds, and lasting 10 seconds.

OTHER OUTCOMES:
Primary Safety Measurement: Serious Adverse Events (SAEs) | 30 days
  We will measure the incidence of all Serious Adverse Events (SAEs)
Secondary Safety Measurement: Adverse Events (AEs): Anticipated and Unanticipated (uAEs) | 30 days
  We will measure the incidence of all Adverse Events (AEs): anticipated and unanticipated (uAEs).

CONTACTS AND LOCATIONS:
Locations (1):
- Assuta HaShalom, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: Undecided